CLINICAL TRIAL: NCT06614751
Title: A Phase I, Open-label, Dose Escalation and Dose Expansion Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Preliminary Efficacy of DAT-2645 in Patients with Advanced/Metastatic Solid Tumors Harboring BRCA1/2 Loss of Function Alterations And/or Other Defects in the DNA Damage Repair Pathway
Brief Title: A PARG Inhibitor DAT-2645 Monotherapy in Patients with Advanced/Metastatic Solid Tumors Harboring BRCA1/2 Loss of Function Alterations And/or Other Defects in the DDR Pathway
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Danatlas Pharmaceuticals Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Danatlas Pharmaceuticals Co.
Record Dates: First submitted 2024-09-18; First posted 2024-09-26 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Solid Cancers; BRCA Mutation; HRD Cancer; Breast Cancer; Prostate Cancer; Colorectal Cancer; Pancreatic Cancer; Endometrial Cancer; Gastric Cancer; Advanced Cancer; Metastatic Solid Tumors
Keywords: PARGi; DAT-2645; PARPi; Advanced solid tumors; Metastatic solid tumors; HRD gene alteration; Homologous recombination; BRCA; BRCA1/2; PALB2; RAD51C; RAD51D
MeSH Terms: conditions — Breast Neoplasms; Prostatic Neoplasms; Colorectal Neoplasms; Pancreatic Neoplasms; Endometrial Neoplasms; Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Part 1, Dose escalation (Experimental): Monotherapy, dose escalation to definite MTD or RDE.
  Interventions: Drug: DAT-2645 tablet
- Module 1 Part 2, Dose optimizing (Experimental): Dose optimizing by 2 dose level after dose escalation to definite RP2D
  Interventions: Drug: DAT-2645 tablet
- Module 2 Part 2, Dose expansion (Experimental): To evaluate safety and efficacy of DAT-2645 tablet in solid tumor under RP2D dosage
  Interventions: Drug: DAT-2645 tablet

INTERVENTIONS:
Drug: DAT-2645 tablet — The patient will be randomized into 2 groups and take DAT-2645 tablet daily. dosage is optimal dose-1 or optimal dose-2, 21day/ Cycle. The subject of this part is to optimize dosage and definite RP2D.
  Arms: Module 1 Part 2, Dose optimizing; Module 2 Part 2, Dose expansion
Drug: DAT-2645 tablet — The study set 6 dose level cohorts in dose escalation part.On C0D1, patient take DAT-2645 one time (Single use), The dosage is same as his enrolled cohort dose level. if no DLT, 7 days later(C1D1), patients will continue taking DAT-2645 tablet daily, dasage is same as before, 21days/cycle.
  Arms: Part 1, Dose escalation

SUMMARY:
The primary objective of the study is to evaluate the safety, tolerability, PK, PD, and prilimary efficacy of a PARG inhibitor DAT-2645 in patients with advanced/metastatic solid tumors harboring BRCA1/2 loss of function alterations and/or other defects in the DNA damage repair (DDR) pathway.

DETAILED DESCRIPTION:
This the the FIH trial of PARG inhibitor DAT-2645.This study will include Part 1 dose escalation study and Part 2 dose expansion study. Eligible patients will be enrolled into Part 1 and Part 2.

In Part 1, 6 dose cohorts will be set and definte MTD/RDE. In Part 2, Dose optimization will be conducted firstly to definite RP2D. dose expansion will be conducted in another 2 cohorts to evaluate the efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent prior to initiation of any procedures in this study.
* At least 18 years of age (inclusive).
* Evidence of an DDR deficiency status in tumor tissue determined by validated testing method.
* Patients with advanced or metastatic solid tumor who have failed standard of care therapy, or are unable to tolerate standard of care therapy, or unable to obtain/unwilling to receive standard therapy. Regardless of PARP inhibitors were used or not in previous treatment.
* At least one measurable lesion by RECIST v1.1 criteria.
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0~2.
* Life expectancy at least 3 months.
* Adequate hematologic and non-hematologic function during the screening.
* Women of childbearing potential must have a negative result of serum pregnancy test at screening.
* Women of childbearing potential or male patients whose spouse have childbearing potential must agree to use a reliable and effective method of contraception during the study and for 6 months after the last dose of the study drug.

Exclusion Criteria:

* Patients who received systemic chemotherapy, small-molecule targeted drugs within 14 days or 5 half-lives (whichever is longer) prior to the first dose of study drug.
* Patients who received biological anti-tumor drugs (including immunotherapy, target therapy, antibody-drug conjugate [ADC]) within 4 weeks prior to the first dose of the study drug.
* Patients who have undergone major surgery within 4 weeks prior to the first dose of study drug.
* Patients who have received radiotherapy within 4 weeks prior to the first dose of study drug (palliative radiotherapy for non-target lesions could be acceptable if it was performed before 14 days prior to the first dose of study drug).
* Any previous treatment with a PARG inhibitor.
* Patients with active CNS metastases (patients with asymptomatic CNS metastases which are imaging stable and not require steroid treatment within 28 days prior to the first dose of study drug, and previous treated breast cancer brain metastasis, can only be enrolled in the Part 2 study).
* Patients who have second primary malignant tumors within the past 3 years prior to screening, except for those who have been cured of basal cell carcinoma, cervical carcinoma in situ, or breast carcinoma in situ.
* Patients with clinically significant cardiovascular or cerebrovascular diseases.
* Active uncontrolled infections requiring intravenous antibiotics or hospitalization.
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of DAT-2645 and no history of bowel obstruction within 6 months prior to enrollment.
* Known pulmonary interstitial disease or pulmonary interstitial fibrosis.
* Patients known hypersensitivity to any component or excipient of DAT-2645.
* Any unresolved toxicities from any prior therapy with severity great than CTCAE Grade 1 prior to start of DAT-2645, except for alopecia and pigmentation and Grade 2 of peripheral sensory neuropathy.
* Participated in other clinical trials (except for screening failure) within 4 weeks prior to the first dose of the study drug in this study.
* Known active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection (active HBV infection is defined as positive hepatitis B surface antigen [HbsAg], or HBV DNA exceeding the lower limit of detection; active HCV infection is defined as positive anti-HCV antibody, and HCV RNA exceeding the lower limit of detection).
* Known human immunodeficiency virus (HIV) infection (patients with adequate CD4+ T cell counts and without history of acquired immune deficiency syndrome [AIDS]-defining opportunistic infections could be enrolled after consultation with sponsor).
* Women who are pregnant or breastfeeding.
* History or evidence of any other clinically significant condition or disease (with the exception of those outlined above) that, in the opinion of the investigator, would be a risk to patient safety or interfere with the study evaluation, procedures or completion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Part 1, Dose esclalation study:To characterize the safety and tolerability of DAT-2645 monotherapy by evaluating the number of participants with dose limiting toxicities, adverse events, and laboratory abnormalities as graded by NCI CTCAE version 5.0 | 6 months
  The incidence of dose limiting toxicites Incidence of treatment-emergent Adverse Events as characterized by type, frequency, severity (as graded by NCI CTCAE version 5.0), timing, seriousness, and relationship to study therapy Laboratory abnormalities as characterized by type, frequency, severity (as graded by NCI CTCAE version 5.0), and timing
Part 2, Dose expansion study: To evaluate preliminary preliminary anti-tumor activity of DAT-2645 tablet monotherapy in participants by measuring tumor Overall Response Rate using RECIST criteria v1.1 | Approximately 2 years
  Tumor response: Overall Response Rate(ORR) assessed by the investigators based on RECIST v1.1 criteria

SECONDARY OUTCOMES:
RP2D | Approximately 6 months
  Recommended Phase 2 dose, will be definite by safety mornitoring committe(SMC).
ORR | Average of 6 months
  Objective Response Rate (ORR) was calculated the rate of response of complete response (CR) or partial response (PR).
DCR | Average of 6 months
  Defined as not meeting the criteria for progression and PR(partial response)
DoR | Approximately 1 years
  DoR(duration of response) per RECIST v1.1(Response Evaluation Criteria in Solid Tumours).
  Measured in CT/MRI image from the time when measurement criteria for complete/ partial response are met till time when progression of the disease is documented.
PFS | Approximately 2 years
  Progression- free survival (PFS) by RECIST V1.1 criteria- from the beginning of treatment to the progression of disease or death.
OS | Approximately 2 years
  Overall Survival (OS) was defined as the time interval between a patient randomized and death from any cause or the end of the last follow-up date.
Area Under the Plasma Concentration Versus Time Curve (AUC) of DAT-2645 | Approximately 1 years
  PK parameters of DAT-2645 and metabolite over time at Cycle 0 Day 1 and at steady state (Cycle 1 Day 21) to model Area Under the the Plasma Concentration Versus Time Curve (AUC) with trough levels at the beginning of every Cycle thereafter
Changes in lysate poly (ADP-ribose) (PAR) level | 6 months
  As a PD parameter, detect the PAR level in peripheral blood mononuclear cell (PBMC) before and after administration of DAT-2645. Explore the correlation between DAT-2645 exposure and PD parameter, safety events.
Correlations between patients' baseline characteristics and effecacy | Approximately 2 years
  Correlations between patients' baseline characteristics (e.g., DDR deficiency type, tumor type) and objective response rate (ORR), to explore the best biomarker for tumor selection.
Time to Achieve Maximal Plasma Concentration (Tmax) of DAT-2645 in Part 1 and Part 2 | Approximately 1 years
  PK parameters of DAT-2645 and metabolite over time at Cycle 0 Day 1 and at steady state (Cycle 1 Day 21) to model time to maximum concentration (Tmax) with trough levels at the beginning of every Cycle thereafter
Maximal Plasma Concentration (Cmax) of DAT-2645 in Part 1 and Part 2 | Approximately 1 years
  PK parameters ofDAT-2645 and metabolite over time at Cycle 0 Day 1-Cycle 0 Day 6 and at steady state (Cycle 1 Day 21) to model maximum concentration (Cmax) with trough levels at the beginning of every Cycle thereafter

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Peking University Cancer Hospital and Institute, Beijing, Beijing Municipality
  - Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijjing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: Yes
only IPD used in the results publication
Supporting Information: Study Protocol, SAP
Time Frame: Danatlas will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please contact with us by information@danatlas.com.
Access Criteria: When a request has been approved Danatlas will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.Please contact with sponsor by email information@danatlas.com